CLINICAL TRIAL: NCT06336447
Title: Can Virtual Reality Improve Patient Tolerance in Patients Undergoing Water Cooled Genicular Nerve Radio Frequency Ablation in Patients With Chronic Knee Pain? A Randomized Controlled Trial
Brief Title: VR and Cooled Genicular Nerve Radio Frequency Ablation for Chronic Knee Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jason Ross, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00220295
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Pain, Chronic
Keywords: Pain; Knee Pain; Virtual Reality; Radio Frequency Ablation; Genicular Nerve Block
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trail.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to study randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group #1: Virtual Reality Headset (Experimental): Group 1 will be assigned to the Virtual Realtity Headset. Participants will wear the headset for at least 10 minutes prior to the planned procedure. Subjects will receive standard procedure. The VR Headset will be removed 10 minutes after the planned procedure.
  Interventions: Other: Experimental: Group #1: Virtual Reality Headset
- Group 2 No Virtual Reality Headset (Active Comparator): Group 2 will receive standard care without the use of the Virtuality Reality Headset.
  Interventions: Other: Group 2 No Virtual Reality Headset

INTERVENTIONS:
Other: Experimental: Group #1: Virtual Reality Headset — Group 1 will be assigned to the Virtual Realtity Headset. Participants will wear the device for at least 10 minutes prior to the planned procedure. Subjects will receive standard procedure. The VR Headset will be removed 10 minutes after the planned procedure.
  Arms: Group #1: Virtual Reality Headset
Other: Group 2 No Virtual Reality Headset — Group 2 will receive standard care without the use of the Virtuality Reality Heaset.
  Arms: Group 2 No Virtual Reality Headset

SUMMARY:
This study will examine the impact of virtual reality used in conjunction with sedation compared to sedation alone in patients undergoing watervcooled genicular nerve ablations for chronic knee pain.

The goals of the study is to determine the relative efficacy of virtual reality as a distraction modality when used as an adjuvant to procedural sedation compared to sedation alone for procedure related pain. To assess procedural satisfaction, and 1-month pain and functional outcomes.To explore whether virtual reality and lower procedure-related pain scores affect 1-month outcomes. And finally to determine whether demographic and clinical characteristics are associated with outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing genicular RFA will be eligible for inclusion in the study
* Patients with knee pain, baseline average of > 4/10
* X-ray evidence of osteoarthritis of the knee
* Pain duration of >6 weeks and no previous knee surgeries
* Patients will also only be included who have never undergone a RFA on the affected knee

Exclusion Criteria:

* Individuals who do not have evidence of osteoarthritis on X-ray,
* Secondary gain expected to influence treatment outcomes
* Poorly controlled psychiatric condition that could affect outcome (e.g. active substance abuse) or impose a barrier to participation
* Chronic opioid use and anticoagulation therapy that cannot be stopped and could warrant a different treatment approach (e.g. phenol ablation)
* Severe motion sickness
* Seizure disorder
* Vision loss
* Pregnant
* Nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Procedural related pain | 10 minutes after procedure
  Reported procedural related pain on a 0-10 verbal rating scale (VRS)

SECONDARY OUTCOMES:
Procedure related satisfaction | 10 minutes after prodedure
  Procedure related satisfaction on a 1-5 Likert scale (5=most satisfied, 1=least satisfied)
Post procedure anxiety | 10 minutes after procedure
  Post-procedural numerical rating scale (NRS) for anxiety on an 11-point scale (0=no anxiety 10=worst possible level of anxiety)
Mean reduction in pain 1 month after procedure | 30 days after procedure
  Mean reduction on a 0-10 numerical rating scale (NRS) pain scores for average and worst knee pain at 1 month
Midazolam administered | 10 minutes before procedure to end of prodedure
  Milligrams of midazolam administered during procedure for sedation
Fentanyl administered | 10 minutes before procedure to end of prodedure
  Micrograms of fentanyl administered during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jason Ross, MD, Principal Investigator — Northwestern Univesity
Locations (1):
- Northwestern Medicine Pain Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Hsu H, Siwiec RM. Knee Osteoarthritis. 2023 Jun 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507884/ PMID 29939661
- [Background] Conger A, Gililland J, Anderson L, Pelt CE, Peters C, McCormick ZL. Genicular Nerve Radiofrequency Ablation for the Treatment of Painful Knee Osteoarthritis: Current Evidence and Future Directions. Pain Med. 2021 Jul 25;22(Suppl 1):S20-S23. doi: 10.1093/pm/pnab129. PMID 34308957
- [Background] Iannaccone F, Dixon S, Kaufman A. A Review of Long-Term Pain Relief after Genicular Nerve Radiofrequency Ablation in Chronic Knee Osteoarthritis. Pain Physician. 2017 Mar;20(3):E437-E444. PMID 28339444
- [Background] Hoffman HG, Richards TL, Van Oostrom T, Coda BA, Jensen MP, Blough DK, Sharar SR. The analgesic effects of opioids and immersive virtual reality distraction: evidence from subjective and functional brain imaging assessments. Anesth Analg. 2007 Dec;105(6):1776-83, table of contents. doi: 10.1213/01.ane.0000270205.45146.db. PMID 18042882
- [Background] Ding J, He Y, Chen L, Zhu B, Cai Q, Chen K, Liu G. Virtual reality distraction decreases pain during daily dressing changes following haemorrhoid surgery. J Int Med Res. 2019 Sep;47(9):4380-4388. doi: 10.1177/0300060519857862. Epub 2019 Jul 25. PMID 31342823
- [Background] Bair MJ, Wu J, Damush TM, Sutherland JM, Kroenke K. Association of depression and anxiety alone and in combination with chronic musculoskeletal pain in primary care patients. Psychosom Med. 2008 Oct;70(8):890-7. doi: 10.1097/PSY.0b013e318185c510. Epub 2008 Sep 16. PMID 18799425